CLINICAL TRIAL: NCT03384953
Title: Chronic Pain Skills Study - Vanderbilt University Medical Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Lindsey Mckernan, Assistant Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170652
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Hypnosis - Group Treatment (Experimental): Subjects will receive 8 weeks of a manualized clinical hypnosis for chronic pain treatment in a group setting. Assessments will be completed before, immediately after, and at 3- and 6- months post-treatment to assess for treatment gains.
  Interventions: Behavioral: Clinical Hypnosis - Group Treatment
- Clinical Hypnosis - Individual Treatment (Experimental): Subjects will receive 8 weeks of a manualized clinical hypnosis for chronic pain treatment in an individual, 1:1 setting. Assessments will be completed before, immediately after, and at 3- and 6- months post-treatment to assess for treatment gains.
  Interventions: Behavioral: Clinical Hypnosis - Individual Treatment

INTERVENTIONS:
Behavioral: Clinical Hypnosis - Group Treatment — group treatment
  Arms: Clinical Hypnosis - Group Treatment
Behavioral: Clinical Hypnosis - Individual Treatment — individual treatment
  Arms: Clinical Hypnosis - Individual Treatment

SUMMARY:
The Osher Center for Integrative Medicine (OCIM) at Vanderbilt is a multidisciplinary outpatient clinic treating patients with chronic pain and complex health issues via integrative services, with goals of improving overall health and wellbeing of those served. At OCIM, clinical hypnosis has been historically provided on an individual basis by the investigator. Due to its impact and increased patient demand for this service, the investigator will be conducting group hypnosis services in addition to individual services order to expand the reach of this program to participants. As such, the investigators see this as a tremendous opportunity to contribute to clinical research to contribute to the evidence based for this form of service by examining participant-reported outcomes associated with completing the treatment. For this project, the investigators seek to assess the impact of a manualized group treatment protocol utilizing clinical hypnosis as a treatment for chronic pain. The investigators will be evaluating participant-reported outcomes to assess the feasibility of conducting hypnosis in this setting, impact of group hypnosis on pain and how participants' responsiveness to hypnosis impacts treatment outcome.

DETAILED DESCRIPTION:
The purpose of this pilot project is to test the efficacy and mechanisms of clinical hypnosis on chronic pain. Primary (characteristic pain intensity) and secondary (mood, quality of life) outcomes will be assessed at pre-treatment, three times during treatment, post-treatment, and at 3- and 6-month follow-up. Potential treatment moderators and mediators will also be assessed. The study will address two aims:

Aim 1: Determine the efficacy of 8 sessions of group delivered HYP training for reducing characteristic pain intensity in patients. The hypothesis associated with Aim 1 is:

Hypothesis 1: Primary Study Hypothesis. Patients receiving 8 sessions of HYP training will report significantly reduced pre- to post-treatment decreases in average pain intensity.

Aim 2 : To evaluate potential moderators (hypnotizability) associated with treatment outcomes following intervention. The hypothesis associated with Aim 2 is:

Hypothesis 2a: Hypnotizability will augment treatment outcomes such that those with higher hypnotizability will experience significantly greater treatment gains.

In addition to testing the above specific hypotheses, we will use the data obtained in this study to further explore (1) the longer-term (up to 6 months) effects of HYP and (2) additional potential moderators (e.g., treatment outcome expectancies, treatment motivation, demographic variables, pain type [neuropathic vs. nociceptive]) and mediators (pain acceptance, catastrophizing, mindfulness, therapeutic alliance, amount of skill practice between sessions) of treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older; *
2. Self-reported presence of chronic pain;**
3. Average pain intensity rating of ≥ 3 on a 0-10 Numerical Rating Scale (NRS) of pain intensity in the last week; **
4. Worst pain intensity rating of ≥ 5 on a 0-10 Numerical Rating Scale (NRS) of pain intensity in the last week;**
5. Duration of chronic pain 3 months or more; **
6. Experiences pain at least 75% of the time in the past 3 months; Those who have a hard time answering this question will be asked the following question: "Which statement best describes your pain?"

   1. Pain all the time, but the pain intensity varies;
   2. Pain most of the time with only occasional periods of being pain-free;
   3. Pain that comes and goes;
   4. Occasional pain; Participants must report experiencing pain that matches one of the first two options;**
7. Able to read, speak, and understand English.**

Exclusion Criteria:

1. Cognitive impairment or limitations (i.e. history of moderate to severe Traumatic Brain Injury (TBI), unresolved TBI, or other medical condition) that would interfere with a patient's ability to participate in a group involving focused attention*.
2. Current or history of diagnosis of primary psychotic or major thought disorder as listed in participant's medical record or self-reported within the past five years;*
3. Hospitalization for psychiatric reasons other than suicidal ideation, homicidal ideation, and/or PTSD self-reported or noted in chart (within the past 5 years);*
4. Psychiatric or behavioral conditions in which symptoms are unstable or severe (e.g. current delirium, mania, psychosis, suicidal ideation, homicidal ideation, substance abuse dependency) as listed in participant's medical record or self-reported within the past six months;*
5. Any behavioral issues as noted in the medical record or by a provider that would indicate the participant may be inappropriate in a group setting;***
6. Presenting symptoms at time of screening that would interfere with participation, specifically active suicidal ideation with intent to harm oneself or active delusional or psychotic thinking;**
7. Difficulties or limitations communicating over the telephone;**
8. Any planned life events that would interfere with participating in the key elements of the study.**
9. Reported average daily use of >120mg morphine equivalent dose (MED). **

   * also verified via medical record review, as described below. **verified solely via self-report, as described below; there is no medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey C McKernan, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Osher Center for Integrative Medicine at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKernan LC, Connors EL, Ryden AM, Finn MTM, Kim A, Vandekar SN, Dmochowski RR, Reynolds WS. Clinical hypnosis can reduce lower urinary tract symptoms in individuals with chronic pain. Neurourol Urodyn. 2023 Jan;42(1):330-339. doi: 10.1002/nau.25090. Epub 2022 Nov 15. PMID 36378832

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clinical Hypnosis - Group Treatment | Clinical Hypnosis - Individual Treatment
Started | 91 | 12
Completed Treatment | 68 | 6
Completed | 51 | 4
Not Completed | 40 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Hypnosis - Group Treatment | Clinical Hypnosis - Individual Treatment | Total
Number analyzed (Participants) | 91 | 12 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.196 (13.894) | 44.833 (13.402) | 50.462 (13.925)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 9 | 74
  Male | 26 | 3 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 75 | 10 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 91 | 12 | 103
Brief Pain Inventory [Mean (Standard Deviation); unit: units on a scale] — Higher values indicate worse pain and possible scale values range from 0 to 10.
  units on a scale | 5.472 (1.736) | 6.125 (1.721) | 5.549 (1.739)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: Brief Pain Inventory (severity scale only) is a 4-item subscale of the Brief Pain Inventory assessing the severity of pain over the past week. Questions inquire into an individual's worst, least, average, and current levels of pain on an 11-point likert scale, with 0 being no pain. It has been validated and is considered the gold standard to utilize in patient-reported outcomes studies. It takes <1 minute to complete.
Time Frame: baseline and 6 months
Population: Patients who completed 6-month post-treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinical Hypnosis - Group Treatment | Clinical Hypnosis - Individual Treatment
Number analyzed (Participants) | 51 | 4
units on a scale | 4.42 (2.173) | 6.625 (1.422)

ADVERSE EVENTS:
Time Frame: 2 months (during 8-session treatment)
Description: In accordance with federal regulations and VUMC policy, adverse events and unanticipated problems involving risk to participants or others that fall under VUMC IRB jurisdiction were reported to the VUMC IRB within 10 working days after learning of the event or problem.
Arm/Group | Clinical Hypnosis - Group Treatment | Clinical Hypnosis - Individual Treatment
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/12
Other Adverse Events (participants affected / at risk) | 0/91 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT03384953/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT03384953/ICF_001.pdf